CLINICAL TRIAL: NCT05895851
Title: Optical Coherence Tomography Angiography Characteristics of Radiation Optic Neuropathy
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-495-01
Record Dates: First submitted 2023-05-18; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Optic Radiation Neuropathy Following Radiotherapy Procedure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RON
  Interventions: Radiation: head and neck radiation
- non-RON: non-RON but with radiiation treatment
  Interventions: Radiation: head and neck radiation
- Normal

INTERVENTIONS:
Radiation: head and neck radiation — RON and non-RON: nasopharyngeal carcinoma patients recieved head and neck radiation; Normal: normal individuals.
  Groups: RON; non-RON

SUMMARY:
Aim: To develop a suitable radiation optic neuropathy (RON) diagnostic model based on optical coherence tomography angiography (OCTA) and to reveal the correlation between endocrine and OCTA indexes in nasopharyngeal carcinoma (NPC) patients with radiation encephalopathy (RE).

Methods: This retrospective cross-sectional study included 80 male NPC patients with RE following radiotherapy (40 non-RON and 40RON). Endocrine and OCTA indexes were collected. The macular and peripapillary vessel density (VD) were automatically analyzed using AngioVue 2.0 of the RTVue XR Avanti device. The OCTA indexes were included in the multivariable binary logistic regression model between non-RON and RON. For all RE patients, a multiple linear regression was performed between each of the OCTA indexes and the endocrine indexes.

DETAILED DESCRIPTION:
Best corrected visual acuity (BCVA) and OCTA (Optovue, Inc., CA, USA) were performed in the RE patients. All examinations were performed by experienced ophthalmic examiners. AngioVue software 2.0 of the RTVue XR Avanti device (Optovue, Inc., CA, USA) was used to perform OCTA imaging. The split-spectrum amplitude-decorrelation angiography (SSADA) algorithm was applied to the scans. Images with a scan quality of not less than 6 were included, while images with obvious artifacts detected by a senior ophthalmologist were excluded. The vessel density (VD) and retinal thickness of the macular and optic nerve head (ONH) area were automatically analyzed in 6 × 6 mm angioretina mode and 4.5 × 4.5 mm angiodisc mode, respectively.

The statistical analyzes were performed using SPSS 24.0 (SPSS Inc., IL, USA). Student's t-test was performed to compare normally distributed variables, while the Mann-Whitney test was performed to compare nonnormally distributed variables. Categorical variables were analyzed with the chi-squared test Statistical significance was set at p < 0.05. The major statistically significant OCTA variables were included in the multivariable binary logistic regression model between NRON and RON. Then, thereceiver operating characteristic (ROC) curve was generated according to the model, and the area under the curve (AUC), sensitivity (SE) and specificity (SP) were reported. In addition, for all RE patients, backward multiple linear regression was performed between each of the above OCTA variables and the statistically significant endocrine indexes.

ELIGIBILITY:
Inclusion Criteria:

(1) Paitients were diagnosed as radiation encephalopathy (RE) confirmed by a neurologist based on magnetic resonance imaging (MRI). The RE patients were divided into RON and non-RON (NRON) groups.

(2）The diagnosis of RON was established according to the following criteria: 1) painless progressive sight loss, 2) abnormal VEP and VF defect, and/or 3) ophthalmoscopic evidence of blurring of the optic disc margins, dilation of retinal veins, hemorrhages, exudates, neovascularization or atrophic optic disc, and/or 4) impaired optic nerve based on MRI.

Exclusion Criteria:

1. other diseases that may cause sight loss, such as stroke, glaucoma, optic neuritis, ischemic optic neuropathy and other optic neuropathy and retinal diseases;
2. NPC recurrence or metastase;
3. uncontrollable diabetes mellitus, hypertension and other serious systemic diseases;
4. lens opacity that affected imaging;
5. an axial length of the included eye greater than 26 mm or a spherical equivalent outside the range between + 3.0 and -3.0 diopters, and
6. a history of intraocular surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The diagnosis of RON was established according to the following criteria: (1) painless progressive sight loss, (2) abnormal VEP and VF defect, and/or (3) ophthalmoscopic evidence of blurring of the optic disc margins, dilation of retinal veins, hemorrhages, exudates, neovascularization or atrophic optic disc, and/or (4) impaired optic nerve based on MRI.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
BCVA | through study completion, an average of 1 year
  best corrected visual acuity

SECONDARY OUTCOMES:
vessel density in the macular area | through study completion, an average of 1 year
vessel density in the ONH area | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zijing Li, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Zijing Li, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No